CLINICAL TRIAL: NCT03764007
Title: 18F-Fluorocholine for the Detection of Parathyroid Adenomas
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Thomas Hope (Other)
Responsible Party: Sponsor-Investigator, Thomas Hope, Associate Professor, Radiology, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-19297
Record Dates: First submitted 2018-11-30; First posted 2018-12-04 (Actual); Results first posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-08

CONDITIONS: Hyperparathyroidism, Primary
Keywords: Positron emission tomography
MeSH Terms: conditions — Hyperparathyroidism, Primary | interventions — fluorocholine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-Fluorocholine PET (Experimental): Patients will undergo a single fluorocholine PET imaging study prior to surgery.
  Interventions: Drug: 18F-Fluorocholine; Procedure: Positron Emission Tomography (PET)

INTERVENTIONS:
Drug: 18F-Fluorocholine — Given intravenously
  Other Names: Fluorocholine
Procedure: Positron Emission Tomography (PET) — Imaging technique that uses radioactive agents known as radiotracers to visualize and measure changes in metabolic processes, and in other physiological activities
  Other Names: PET

SUMMARY:
The investigators are studying the ability of F18 labeled fluorocholine PET to localize parathyroid adenomas in patients with hyperparathyroidism prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Biochemically proven hyperparathyroidism and an indication for surgery
* Age >= 13 years old
* Karnofsky performance status of > 50 (or Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) equivalent).
* Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

* Patients exceeding the weight limitations of the scanner or are not able to enter the bore of the PET scanner due to BMI.
* Inability to lie still for the entire imaging time (e.g. cough, severe arthritis, etc.).
* Inability to complete the needed investigational due to other reasons (severe claustrophobia, radiation phobia, etc.).
* Pregnancy.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hope, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Journal of Nuclear Medicine, published on March 5, 2021 as doi:10.2967/jnumed.120.256735 — https://jnm.snmjournals.org/content/early/2021/03/12/jnumed.120.256735

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 18F-Fluorocholine PET
Started | 98
Imaging Completed | 98
Underwent Parathyroidectomy Surgery | 77
Completed | 77
Not Completed | 21

BASELINE CHARACTERISTICS:
Arm/Group | 18F-Fluorocholine PET
Number analyzed (Participants) | 98
Age, Continuous [Median (Full Range); unit: years] | 64 [17 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 83
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 64
  More than one race | 5
  Unknown or Not Reported | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 98
Prior History of Parathyroidectomy at Baseline [Count of Participants; unit: Participants] | 41

OUTCOME MEASURES:

1. Primary Outcome: Proportion of True Positives for the Overall Detection of the Abnormal Parathyroid Adenoma
Description: The true positive (sensitivity) rate is defined as the proportion of participants with location of the suspected adenoma on 18F-Fluorocholine PET correlating with location of an abnormal parathyroid at time of participant surgery. For a patient with multiple hyperplastic glands, only one gland needs to correlate for the patient to count as a true positive. For analysis, adenomas described as arising in the mid thyroid bed will considered correct if located in either the inferior or superior bed. Patients will be followed-up to determine if they undergo a parathyroidectomy for up to 1 year.
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 18F-Fluorocholine PET
Number analyzed (Participants) | 77
proportion of participants | 0.75 [0.63 to 0.82]

2. Primary Outcome: Proportion of True Positives for the Detection of the Abnormal Parathyroid Adenoma Using Sestamibi Imaging
Description: The true positive (sensitivity) rate is defined as the proportion of participants with location of the suspected adenoma on 18F-Fluorocholine PET correlating with location of an abnormal parathyroid at time of participant surgery. For a patient with multiple hyperplastic glands, only one gland needs to correlate for the patient to count as a true positive. In patients who had a sestamibi study performed prior to the fluorocholine imaging study, the original dictated report from the sestamibi will be used for comparison. For analysis, adenomas described as arising in the mid thyroid bed will considered correct if located in either the inferior or superior bed. Patients will be followed-up to determine if they undergo a parathyroidectomy for up to 1 year.
Time Frame: Up to 1 year
Population: Only 66 of the 77 participants who underwent surgery had an available sestamibi study
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 18F-Fluorocholine PET
Number analyzed (Participants) | 66
proportion of participants | 0.70 [0.59 to 0.79]

3. Secondary Outcome: Detection Rate in Patients Who Have Not Undergone Surgical Resection
Description: The detection rate is defined as the proportion of participants with a 18F-fluorocholine PET positive read who do not subsequently undergo parathyroidectomy, using the dictated reports to determine the detection sensitivity for parathyroid adenomas. Patients will be followed-up to determine if they undergo a parathyroidectomy for up to 1 year.
Time Frame: Up to 1 year
Measure: Number; unit: proportion of participants
Arm/Group | 18F-Fluorocholine PET
Number analyzed (Participants) | 21
proportion of participants | 0.90

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | 18F-Fluorocholine PET
All-Cause Mortality (participants affected / at risk) | 0/98
Serious Adverse Events (participants affected / at risk) | 0/98
Other Adverse Events (participants affected / at risk) | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT03764007/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-04): https://cdn.clinicaltrials.gov/large-docs/07/NCT03764007/ICF_001.pdf